CLINICAL TRIAL: NCT03643484
Title: IMFINZI® Injection 120 mg, 500 mg Specific-Clinical Experience Investigation in Patients With Locally Advanced Unresectable Non-small Cell Lung Cancer Who Are Treated With Maintenance Therapy After Definitive Chemoradiation Therapy.
Brief Title: IMFINZI Specific-Clinical Experience Investigation in Patients With NSCLC After Definitive Chemoradiation Therapy
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4194C00003
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung Diseases, Interstitial; Radiation Pneumonitis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Diseases, Interstitial; Radiation Pneumonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

SUMMARY:
To investigate the impact of presence/absence or grade of radiation pneumonitis before starting IMFINZI, on the onset of interstitial lung disease (including radiation pneumonitis) after starting IMFINZI, in the real world in patients with locally advanced unresectable non-small cell lung cancer who are treated with the product as maintenance therapy after definitive chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

-Patients with locally advanced unresectable non-small cell lung cancer who are treated with IMFINZI for the first time as maintenance therapy after definitive chemoradiation therapy

Exclusion Criteria:

-No past history of hypersensitivity to the components of IMFINZI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally advanced unresectable non-small cell lung cancer after definitive chemoradiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Interstitial lung disease (including radiation pneumonitis) by post-chemoradiation therapy radiation pneumonitis (yes/no) and by severity (CTCAE grade) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (36):
- Japan (36):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4194C00003&attachmentIdentifier=e524dac4-f399-4aec-8624-e98223e53e3c&fileName=D4194C00003__Final_report.pdf&versionIdentifier=